CLINICAL TRIAL: NCT03071341
Title: An Extension Study Evaluating Long Term Safety and Activity of AGT-181 in Patients With Mucopolysaccharidosis I Who Were Previously Enrolled in Studies With AGT-181
Brief Title: Extension Study Evaluating Long Term Safety and Activity of AGT-181 in Children With MPS I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ArmaGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGT-181-101E
Record Dates: First submitted 2017-02-27; First posted 2017-03-06 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Mucopolysaccharidosis I
Keywords: MPS I; Hurler Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — valanafusp alpha

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to 1.0, 3.0 or 6.0 mg/kg (same dose taken during the previous study, AGT-181-101)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AGT-181 (Experimental): Human Insulin Receptor Monoclonal Antibody-Human alpha-L-iduronidase (HIRMAb-IDUA) fusion protein
  Interventions: Drug: AGT-181

INTERVENTIONS:
Drug: AGT-181 — Human Insulin Receptor Monoclonal Antibody-Human alpha-L-iduronidase (HIRMAb-IDUA) Fusion Protein

SUMMARY:
AGT-181 is a fusion protein containing alpha-L-iduronidase that is intended to deliver the enzyme peripherally and to the brain, when administered intravenously.

This is a long term safety and tolerability study of AGT-181 in patients with MPS I who completed the previous 26-week study, AGT-181-101. Information on the biological activity of the investigational drug will also be collected.

DETAILED DESCRIPTION:
AGT-181-101E is a safety and tolerability study of AGT-181 in patients with MPS I who completed the previous 26-week study, AGT-181-101. Information on the biological activity of the investigational drug will be collected as well as longitudinal safety information.

ELIGIBILITY:
Inclusion Criteria:

* 2 years of age or older (and less than 18)
* Must have been previously enrolled in study AGT-181-101
* Written consent and assent as required
* Female patients must not be pregnant, willing to utilize appropriate birth control methods and undergo pregnancy testing during the study

Exclusion Criteria:

* Refusal to complete all assessments
* Pregnant or Lactating
* Received investigational drug within 1 year prior to study enrollment
* Medical condition or extenuating circumstance that, in the opinion of the investigator, may interfere with study compliance
* Clinically significant spinal cord compression or evidence of cervical instability (i.e. expected to require intervention during study participation)
* Has developed clinically relevant hypersensitivity/anaphylactoid reactions to AGT-181

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events as a measure of safety and tolerability | 24 months
  Incidence and prevalence of adverse events

SECONDARY OUTCOMES:
Total urinary glycosaminoglycans (GAGs) | 24 months
  Change in total urinary glycosaminoglycans (GAGs)
Urinary heparan sulfate and dermatan sulfate | 24 months
  Change in urinary heparan sulfate and dermatan sulfate
Plasma heparan sulfate and dermatan sulfate | 24 months
  Change in plasma heparan sulfate and dermatan sulfate
CSF heparan sulfate and dermatan sulfate | 24 months
  Change in CSF heparan sulfate and dermatan sulfate
liver and/or spleen volume | 24 months
  Change in liver and/or spleen volume measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P Rioux, MD PhD, Study Director — ArmaGen, Inc
Locations (1):
- HCPA - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giugliani R, Giugliani L, de Oliveira Poswar F, Donis KC, Corte AD, Schmidt M, Boado RJ, Nestrasil I, Nguyen C, Chen S, Pardridge WM. Neurocognitive and somatic stabilization in pediatric patients with severe Mucopolysaccharidosis Type I after 52 weeks of intravenous brain-penetrating insulin receptor antibody-iduronidase fusion protein (valanafusp alpha): an open label phase 1-2 trial. Orphanet J Rare Dis. 2018 Jul 5;13(1):110. doi: 10.1186/s13023-018-0849-8. PMID 29976218